CLINICAL TRIAL: NCT00563251
Title: Azithromycin Therapy for Bronchiolitis Obliterans Syndrome After Allogenic Bone Marrow Transplantation
Brief Title: Effectiveness of Azithromycin Therapy in Improvement of Symptoms and Lung Function in Patients With Bronchiolitis Obliterans After Bone Marrow Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: The University of Hong Kong (Other); Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 04-165 T/487; HARECCTR0500038
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Bronchiolitis Obliterans; Bone Marrow Transplantation
Keywords: Bronchiolitis obliterans in bone marrow transplant recipients
MeSH Terms: conditions — Bronchiolitis Obliterans | interventions — Azithromycin

INTERVENTIONS:
Drug: Azithromycin
Drug: Placebo tablet

SUMMARY:
Bronchiolitis obliterans syndrome (BOS), an obstructive airway disease as a result of chronic rejection, is one of the major causes of morbidity and mortality in long-term survivors of allogeneic bone marrow transplantation (BMT). Although augmentation of immunosuppressive treatment might help but the only effective treatment for BOS is by lung transplantation.

Macrolide antibiotics, which have been licensed to use as antibacterial agents for decades, have been found to have immunomodulatory properties in addition to their antibacterial activity. Low dose Azithromycin, an antibiotic of the macrolide family, has been shown to have promising result in a pilot study in treating BOS associated with lung transplantation. We propose to perform a prospective, randomised, double blind study to test the efficacy of Azithromycin in treating BOS after BMT. Patients with proven BOS after BMT will be randomised into two groups based on lung function parameters. One group will receive low dose Azithromycin while placebo will be provided for the other group. Lung function will be serially monitored at 3 month, 6 months and 12 months after commencement of treatment with drug/placebo. If Azithromycin was proven effective in treating BOS then all patient with proven BOS should be treated with this drug.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed BOS post BMT
* Informed consent

Exclusion Criteria:

* Women currently pregnant or nursing
* Allergy to macrolide

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-04; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Quality of life assessment by questionnaires | 3 months after treatment
Spirometry | 3 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Albert Lie, Dr, Principal Investigator — Department of Medicine, Queen Mary Hospital/ The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China